CLINICAL TRIAL: NCT00018421
Title: Effects of Exercise on Patients With Hemiparetic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: CADE-RA
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Stroke; Hemiplegia; Cardiovascular Disease
Keywords: Cerebrovascular Disorders; Exercise; Rehabilitation
MeSH Terms: conditions — Stroke; Hemiplegia; Cardiovascular Diseases; Cerebrovascular Disorders; Motor Activity

INTERVENTIONS:
Procedure: Treadmill Exercise

SUMMARY:
This randomized trial investigates the hypothesis that regular aerobic exercise training using a task specific gait training modality will improve cardiovascular fitness, functional mobility, and reduce risk factors for recurrent cardiovascular events in chronic hemiparetic stroke patients, when compared to matched controls performing just stretching.

DETAILED DESCRIPTION:
The aims are to determine whether 6 months progressive graded treadmill training: 1) improves cardiovascular fitness levels and reduces the excessive energy demands of hemiparetic gait, as defined by oxygen consumption levels based on open circuit spirometry during peak and submaximal exercise ambulation tasks; 2) increases free living physical activity measured by portable kinematic recording devices and quantitative in vivo determination of energy expenditure using stable isotopes; and, 3) improves the cardiovascular-metabolic risk factor profile including measures of key endogenous fibrinolysis regulatory enzymes [plasma tissue plasminogen activator (t-PA) and its main circulating inhibitor (PAI-1)], fasting lipoprotein lipid profiles, blood pressure, and oral glucose tolerance and insulin responses. Measurements of body composition at baseline and after training will further determine the effects of aerobic exercise training on muscle mass and central obesity.

ELIGIBILITY:
Males or Females Ages 40 yrs to 80 yrs who are chronic hemiparetic stroke patients.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-07; Study Completion 2001-06

CONTACTS AND LOCATIONS:
Locations (1):
- VA Maryland Health Care System, Baltimore, Maryland, United States